CLINICAL TRIAL: NCT01450462
Title: Vitamin D and Sexual Health (the DASH Study)
Brief Title: Vitamin D and Sexual Health
Acronym: DASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Abigail Norris Turner, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: KL2RR025754-ANT; KL2RR025754 (NIH)
Record Dates: First submitted 2011-10-07; First posted 2011-10-12 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (cholecalciferol) (Experimental)
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol)
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (cholecalciferol) — Women in the vitamin D arm take 50,000 international units (IU) of vitamin D3 (cholecalciferol) weekly for four weeks (end of week 1, week 2, week 3 and week 4), then every 4 weeks through 24 weeks of follow-up (end of week 8, week 12, week 16, week 20 and week 24) for a total of 9 treatments
  Arms: Vitamin D (cholecalciferol)
Dietary Supplement: Placebo — Women in the placebo arm will take their matching supplement weekly for four weeks (end of week 1, week 2, week 3 and week 4), then every 4 weeks through 24 weeks of follow-up (end of week 8, week 12, week 16, week 20 and week 24) for a total of 9 treatments
  Arms: Placebo

SUMMARY:
Bacterial vaginosis (BV) develops when the concentration of healthy Lactobacillus species in the vagina declines and is replaced by other bacterial species. BV is the most common vaginal infection worldwide, but the etiology of this complex condition is not clear. BV is associated with a 60% increased risk of HIV acquisition as well as numerous other detrimental reproductive outcomes. A profound racial disparity exists in BV prevalence in women in the United States (US): 23% of white women versus. 52% of black women have BV. The investigators hypothesize that inadequate vitamin D contributes to BV development and/or recurrence. Vitamin D is essential to immune function, serving both to stimulate mechanisms associated with pathogen elimination and to regulate immune response. According to nationally-representative data, 90% of US blacks have insufficient vitamin D levels. In two recent analyses, low vitamin D was associated with higher BV prevalence in pregnant African-Americans; a third replicated this finding in pregnant African-American and white women. The investigators wish to conduct a small, pilot randomized controlled trial (RCT) to assess the effect of vitamin D supplementation among non-pregnant, BV-positive women at a public sexually transmitted disease (STD) clinic. This small (n=150), two-arm, placebo-controlled, masked, 24-week RCT of high-dose vitamin D supplementation will inform the development of future large-scale RCT design and implementation.

ELIGIBILITY:
Inclusion Criteria:

* speak English;
* be between 18 and 50 years old, inclusive;
* be pre-menopausal;
* have at least one ovary;
* be positive for bacterial vaginosis

Exclusion Criteria:

* pregnant at enrollment or in the previous 3 months;
* planning to become pregnant in the next six months;
* currently breastfeeding;
* currently be menstruating heavily;
* have a contraindication to oral metronidazole treatment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Serum vitamin D level | 24 weeks
  To assess the effect of vitamin D supplementation on serum vitamin D levels after 24 weeks
Serum and cervical immunoinflammatory mediators | 24 weeks
  To assess the effect of vitamin D supplementation on levels of and correlations between BV-associated and vitamin D-associated immunoinflammatory mediators after 24 weeks
Bacterial vaginosis recurrence | 24 weeks
  To assess the effect of high-dose vitamin D on recurrence of bacterial vaginosis

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Norris Turner, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Columbus Public Health Sexual Health Clinic, Columbus, Ohio, United States

REFERENCES:
- [Derived] Turner AN, Carr Reese P, Fields KS, Anderson J, Ervin M, Davis JA, Fichorova RN, Roberts MW, Klebanoff MA, Jackson RD. A blinded, randomized controlled trial of high-dose vitamin D supplementation to reduce recurrence of bacterial vaginosis. Am J Obstet Gynecol. 2014 Nov;211(5):479.e1-479.e13. doi: 10.1016/j.ajog.2014.06.023. Epub 2014 Jun 17. PMID 24949544